CLINICAL TRIAL: NCT01077583
Title: Performance Evaluation Study for Clearblue Pregnancy Test
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-0148
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-01

CONDITIONS: Pregnancy
Keywords: Pregnancy test; Wishing to become pregnant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Daily early morning urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect urine samples and dating scan information from women who wish to become pregnant. Urine samples will be tested in the laboratory with the Clearblue Pregnancy Test and the results correlated with volunteer information.

DETAILED DESCRIPTION:
Approximately 800 female volunteers wishing to become pregnant will be recruited locally around 5 trial centers within the US.

Daily urine samples and gestational age dating scan information obtained from the study will be used in laboratory tests to assess the accuracy of the Clearblue Pregnancy Test. Product assessment will involve testing of early morning urine samples collected by women during the cycle in which they conceived. Urine samples will be collected pre-conception to the end of the second trimester.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study and agree to comply with study procedures.
* Has menstrual bleeds.
* Seeking to become pregnant.
* Intend to seek medical care during pregnancy.

Exclusion Criteria:

* Has positive pregnancy test on screening.
* Has received medical treatment for infertility or is participating in an assisted fertility program.
* Known condition to contra-indicate pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligibility:
  Ages Eligible for study: 18 - 45 years. Gender Eligible for study Female. Healthy Volunteers Yes.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The agreement of the Clearblue Pregnancy Test result with Duration of Pregnancy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Marx, MD, Principal Investigator — Radiant Research
Locations (5):
- United States (5):
  - Radiant Research Inc, Atlanta, Georgia
  - Radiant Research, Inc., Chicago, Illinois
  - Radiant Research Inc, Edina, Minnesota
  - Radiant Research Inc, Dallas, Texas
  - Radiant Research Inc, San Antonio, Texas

REFERENCES:
- [Derived] Larsen J, Buchanan P, Johnson S, Godbert S, Zinaman M. Human chorionic gonadotropin as a measure of pregnancy duration. Int J Gynaecol Obstet. 2013 Dec;123(3):189-95. doi: 10.1016/j.ijgo.2013.05.028. Epub 2013 Sep 3. PMID 24079475